CLINICAL TRIAL: NCT04706091
Title: Efficacy of Suvorexant in Patients With Effectively Treated Restless Legs Syndrome and Persistent Chronic Insomnia: A Randomized Placebo-Controlled Crossover Trial
Brief Title: Efficacy of Suvorexant in Patients With Effectively Treated Restless Legs Syndrome and Persistent Chronic Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, John Winkelman, MD, PhD, Chief, Sleep Disorders Clinical Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P003535
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-12

CONDITIONS: Restless Legs Syndrome; Insomnia; Sleep Disorder
Keywords: Suvorexant
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to suvorexant 10-20 mg or equivalent placebo for four weeks followed by crossover (after a 2-week washout) to the alternate treatment.
Who Masked: Participant, Investigator
Masking Description: The participant, investigator, and clinical research coordinator will remain masked throughout the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment --> Placebo (Experimental): This group will receive suvorexant during the first 4-week phase, and placebo during the second 4-week phase.
  Interventions: Drug: Suvorexant; Other: Placebo
- Placebo --> Treatment (Experimental): This group will receive placebo during the first 4-week phase, and suvorexant during the second 4-week phase.
  Interventions: Drug: Suvorexant; Other: Placebo

INTERVENTIONS:
Drug: Suvorexant — 10-mg or 20-mg suvorexant capsules
  Other Names: Belsomra
Other: Placebo — Matching placebo capsules

SUMMARY:
The investigators aim to determine the effect of suvorexant on actigraphically-derived total sleep time in patients with effectively treated restless legs syndrome with persistent insomnia in a two-arm, double-blind, randomized placebo-controlled crossover 2.5-month trial.

DETAILED DESCRIPTION:
Restless Legs Syndrome (RLS) is a sensory-motor neurological disorder characterized by an irresistible urge to move the legs. Persistent difficulties with all phases of sleep are common in patients whose RLS symptoms are resolved with treatment. Multiple potential causes for treatment-refractory sleep disturbance exist, including activating effects of dopamine agonists (which are first-line RLS treatments), conditioned insomnia and poor sleep habits as a result of chronic RLS-related sleep disturbance, and comorbid medical and psychiatric illness. Suvorexant provides an important therapeutic option to treat insomnia in the context of RLS. It has demonstrated long-term efficacy, particularly in shortening the duration of nocturnal awakenings and increasing total sleep time. Similarly, it has a comparatively benign side effect profile compared to many other agents typically prescribed to treat insomnia. The investigators aim to determine the effect of suvorexant on actigraphically-derived total sleep time, as well as actigraphically-derived wake after sleep onset, Insomnia Severity Index score, subjective sleep endpoints, and RLS symptom severity.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of any ethnic origin
2. Written informed consent is obtained
3. Speaks and writes in English
4. A willingness and ability to comply with study procedures
5. Age 25-85 years
6. Diagnosis of RLS via Cambridge-Hopkins RLS questionnaire
7. International Restless Legs Syndrome Study Group scale score (IRLS) < 15
8. RLS treatment with a dopaminergic agonist or an alpha-2-delta agent
9. No changes in RLS medication in the previous month
10. DSM-5 criteria for Insomnia Disorder
11. Report a total sleep time ≤ 7 hours and wake after sleep onset (WASO) > 45 minutes on 7 or more of the 14 nightly sleep logs during both the initial 2-week screening period and the two-week screening run-in period. WASO does not decrease by more than 50% on the 2-week sleep diary obtained between the screening visit and the randomization visit

Exclusion Criteria:

1. Diagnosis of moderate/severe obstructive sleep apnea (AHI > 30) not using continuous positive airway pressure therapy (CPAP) (can be included if CPAP adherent), or other untreated primary sleep disorders (e.g. narcolepsy)
2. Shift workers
3. Unwillingness to not use sedative-hypnotics (other than suvorexant) during the study period
4. Unwillingness to maintain stable RLS medication during the study unless medically indicated
5. Current use of an opiate medication
6. Unwillingness to not take stimulants (e.g. caffeine) after 4:00 pm during the study
7. Current major depressive episode, by report and as indicated by the Patient Health Questionnaire (PHQ-9)
8. Lifetime history of bipolar disorder, psychosis, or other serious psychiatric illness
9. Current alcohol/substance use disorder
10. BMI ≥ 40 kg/m^2
11. Renal or hepatic disease judged to interfere with drug metabolism and excretion
12. Pregnancy or breastfeeding
13. Malignancy within past 2 years
14. Surgery within past 3 months
15. Neurological disorder or cardiovascular disease raising safety concerns about use of suvorexant and/or judged to interfere with ability to assess efficacy of the treatment
16. Medical instability considered to interfere with study procedures
17. Concomitant medications with drug interaction or co-administration concerns
18. Contraindications or allergic responses to suvorexant
19. History of being treated with suvorexant
20. Travel across two time-zones during the week prior to enrollment
21. Greater than 6 cups of coffee per day

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Winkelman, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winkelman JW, Zackon J, Kilty A. Improvement in self-reported, but not actigraphic, sleep measures with suvorexant in people with well-controlled Restless Legs Syndrome and persistent insomnia. Sleep Med. 2024 Dec;124:30-37. doi: 10.1016/j.sleep.2024.09.005. Epub 2024 Sep 8. PMID 39260076

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to signing an Informed Consent Form (ICF), participants complete Sleep Diaries. If eligible, they sign the ICF, followed by additional Sleep Diaries. During this second period, 8 enrolled participants were excluded from the study for the following reasons: sleep no longer met criteria (4), RLS was too severe (2), sleep apnea (1), no RLS (1). Four participants withdrew from the study due to: unrelated surgery (2), no longer interested (1), lost to follow-up (1).
Period: Treatment 1
Arm/Group | Treatment --> Placebo | Placebo --> Treatment
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0
Period: Treatment 2
Arm/Group | Treatment --> Placebo | Placebo --> Treatment
Started (One participant in the Treatment --> Placebo group withdrew before treatment period 2 due to starting CBT.) | 17 | 16
Completed | 16 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment --> Placebo | Placebo --> Treatment | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (7.7) | 59.3 (10.9) | 62.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 16 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 16 | 34
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (10.1) | 27.0 (4.8) | 28.1 (8.0)
International Restless Legs Syndrome Study Group Rating Scale (IRLS) [Mean (Standard Deviation); unit: units on a scale (0-40)] — The International Restless Legs Syndrome Study Group Rating Scale (IRLS) is a questionnaire that measures Restless Legs Syndrome symptom severity on a scale from 0-40, 40 representing the most severe and frequent symptoms, and 0 being the least.
  units on a scale (0-40) | 8.3 (5.9) | 8.1 (4.5) | 8.2 (5.2)
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale (0-28)] — The Insomnia Severity Index (ISI) is a questionnaire that measures insomnia severity on a scale from 0-28, 28 representing severe clinical insomnia and 0 representing no clinical insomnia.
  units on a scale (0-28) | 16 (3.9) | 14.2 (3.8) | 15.1 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Actigraphically-Derived Total Sleep Time
Description: Change in mean total sleep time (between baseline and end of treatment, for each treatment period), as measured by actigraphy. Participants wear an actigraph watch, which assesses periods of activity and rest to determine the total amount of sleep during one sleep period. Total sleep time excludes sleep onset latency and nighttime awakenings.
Time Frame: 2 weeks
Population: Two participants in the Treatment --> Placebo arm of the study withdrew prior to treatment period 2.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment --> Placebo | Placebo --> Treatment
Number analyzed (Participants) | 18 | 16
Minutes
  Treatment 1 | 5.03 (40.80) | 11.44 (24.16)
  Treatment 2: number analyzed (Participants) | 16 | 16
  Treatment 2 | 7.60 (53.01) | 17.96 (32.04)

2. Secondary Outcome: Actigraphically-Derived Wake After Sleep Onset
Description: Change in wake after sleep onset (between baseline and end of treatment, for each treatment period), as measured by actigraphy. Participants wear an actigraph watch, which assesses periods of activity and rest to determine the total wake time after sleep onset, during nighttime awakenings.
Time Frame: 2 weeks
Population: Two participants in the Treatment --> Placebo arm withdrew from the study prior to treatment period 2.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment --> Placebo | Placebo --> Treatment
Number analyzed (Participants) | 18 | 16
Minutes
  Treatment 1 | 0.88 (14.26) | -0.67 (19.53)
  Treatment 2: number analyzed (Participants) | 16 | 16
  Treatment 2 | -1.05 (15.59) | -1.20 (12.05)

3. Secondary Outcome: Insomnia Severity Index
Description: Change in ISI score between baseline and end of treatment, for each treatment period. The ISI is a validated tool to measure insomnia severity, on a scale of 0-28, with a higher score representing greater insomnia severity.
Time Frame: 2 weeks
Population: Two participants in the Treatment --> Placebo arm withdrew from the study prior to treatment period 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment --> Placebo | Placebo --> Treatment
Number analyzed (Participants) | 18 | 16
units on a scale
  Treatment 1 | -4.78 (4.62) | -1.25 (5.30)
  Treatment 2: number analyzed (Participants) | 16 | 16
  Treatment 2 | -4.29 (5.30) | -5.69 (6.87)

ADVERSE EVENTS:
Time Frame: AE data were collected during the two treatment periods, for a total of 8 weeks.
Groups:
- Suvorexant: Participants in both arms of the study received suvorexant treatment, either during treatment one or treatment two.
- Placebo: Participants in both arms of the study received placebo treatment, either during treatment one or treatment two.
Arm/Group | Suvorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 18/34 | 12/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Suvorexant (N=34) | Placebo (N=32)
Fatigue (General disorders) | 10 | 3
Vivid Dreams (Psychiatric disorders) | 3 | 1
Worsened RLS (Nervous system disorders) | 3 | 6
Headache (General disorders) | 2 | 4
Mood Alteration (Depression/Anxiety/Irritability) (Psychiatric disorders) | 2 | 3
Worsened Insomnia (Psychiatric disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT04706091/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT04706091/ICF_001.pdf